CLINICAL TRIAL: NCT05910411
Title: Inelastic Compression in Edema After Revascularization
Acronym: COMPRIME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-AOIP-02; 2022-A02260-43 (Registry Identifier: ANSM)
Record Dates: First submitted 2023-06-02; First posted 2023-06-18 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Inelastic compression (Experimental): Inelastic compression used in the treatment of lymphedema
  Interventions: Device: Inelastic compression

INTERVENTIONS:
Device: Inelastic compression — Inelastic compression used in the treatment of lymphedema

SUMMARY:
The appearance of revascularization edema of the lower limb is a frequent complication in peripheral vascular surgery. It can lead to a delay in healing and even to trophic disorders.

The prevention and treatment of this complication have so far been limited to postural measures (elevation of the limbs), in the absence of other recommendations and given the contraindication of elastic compression.

Inelastic compression is another mode of compression sometimes used in the treatment of lymphedema. It exerts a stable continuous pressure regardless of the patient's position. The investigator's aim is to demonstrate that compression with inelastic bands, applied under good conditions, does not have a major effect on distal arterial vascularization in arterial patients who have undergone revascularization by supra-articular bypass or endovascular treatment of the lower limb.

ELIGIBILITY:
Inclusion Criteria:

1. patients over 18 years of age
2. arteriopathic patients requiring femoropopliteal revascularization by bypass surgery who have been revascularized
3. signature of an informed consent
4. person affiliated or beneficiary of a social security plan

Exclusion Criteria:

1. arterial bypasses under the leg or distal joints
2. critical ischemia
3. patients operated on for acute ischemia
4. pregnant or breast-feeding women
5. severe cardiac insufficiency

5) severe peripheral neuropathy 6) allergies to the components of the tapes 7) persons deprived of liberty by judicial or administrative decision 8) persons under legal protection

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-11 (Estimated)

PRIMARY OUTCOMES:
Evaluating the safety of inelastic compression | day 5
  no skin complications OR a drop in toe blood pressure and/or transcutaneous oxygen pressure (TCPO2) and/or TMS of 20% before and after placement of the compression

SECONDARY OUTCOMES:
threshold of cPSI below which the application of inelastic compression results in altered arterial flow. | day 5
  Determine the threshold of IPSc values before and after compression placement
toe pressure below which the application of inelastic compression results in altered arterial flow. | day 5
  Determine the toe pressure based on TCPO2 values before and after compression placement

CONTACTS AND LOCATIONS:
Overall Officials: PASCAL GIORDANA, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France, France

IPD SHARING:
Plan to Share IPD: No